CLINICAL TRIAL: NCT01138046
Title: An Open-label, Single-arm, Phase I/II Study of Lapatinib in Combination With Weekly Paclitaxel as First-line Chemotherapy for ErbB2-overexpressing Metastatic Breast Cancer Patients
Brief Title: Phase I/II Study of Lapatinib in Combination With Paclitaxel as 1L Chemotherapy for ErbB2-positive MBC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 113806
Record Dates: First submitted 2010-03-18; First posted 2010-06-07 (Estimated); Results first posted 2014-09-19 (Estimated); Last update posted 2014-10-07 (Estimated); Status verified 2014-09

CONDITIONS: Neoplasms, Breast
Keywords: advanced/metastatic breast cancer; lapatinib; ErbB2; ErbB2-overexpressing; pharmacokinetics; dual kinase inhibitor; HER-2/neu; EGFR; ErbB1
MeSH Terms: conditions — Breast Neoplasms | interventions — Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lap+weekly Pacli (Experimental): These subjects will receive weekly paclitaxel (80 mg/m2 IV for 3 weeks in a 4 week cycle) plus lapatinib. Subjects will receive a daily dose of lapatinib until disease progression or withdrawal from study treatment due to unacceptable toxicity or withdrawal of consent.
  Interventions: Drug: Lapatinib in combination with weekly paclitaxel

INTERVENTIONS:
Drug: Lapatinib in combination with weekly paclitaxel — These subjects will receive weekly paclitaxel (80 mg/m2 IV for 3 weeks in a 4 week cycle) plus lapatinib (1500 mg once daily, starting on the second day of phase I). Subjects will receive a daily dose of lapatinib until disease progression or withdrawal from study treatment due to unacceptable toxicity or withdrawal of consent. Study completion is defined as deaths after administering study treatment for more than once. Subjects will be treated with paclitaxel for standard of 6 cycles, and may be continued at the discretion of investigators. If the subject experiences progression, an unacceptable toxicity related to paclitaxel, or termination of lapatinib therapy, paclitaxel therapy must be terminated any time of study period, even before 6 cycles of paclitaxel are given.

SUMMARY:
This is an open-label, non-randomized, multi-center study of lapatinib plus paclitaxel to evaluate safety, tolerability and efficacy in Japanese patients with ErbB2 over expressing advanced or metastatic breast cancer. Lapatinib 1500mg/day will be administered in combination with paclitaxel 80mg/m2/week. Lapatinib and paclitaxel will be administered until disease progression or withdrawal from the study due to unacceptable toxicity.

The study will proceed in two phases. The first phase (Phase I part) will lead to evaluate safety and tolerability of lapatinib taken together with paclitaxel in the first 6 subjects. Pharmacokinetic profile also will be evaluated as the secondary objects.

Then the study will move to the next treatment phase (Phase II part) to evaluate further safety and clinical activity, if no major safety concerns are raised during Phase I part. The primary objective of the study is to evaluate overall survival (OS), and the secondary objectives are Objective tumour response rate (ORR), Duration of response, Time to response, Clinical benefit and Progression-free survival (PFS) in 12 subjects.

DETAILED DESCRIPTION:
This is an open-label, single-arm, Phase I/II study to evaluate the efficacy, safety and tolerability of weekly paclitaxel and lapatinib in subjects with ErbB2-overexpressing advanced or metastatic breast cancer who have not received prior therapy for metastatic disease. These subjects will receive weekly paclitaxel (80 mg/m2 IV for 3 weeks in a 4 week cycle) plus lapatinib (1500 mg once daily). Subjects will receive a daily dose of lapatinib until disease progression or withdrawal from study treatment due to unacceptable toxicity or withdrawal of consent. Subjects will be treated with paclitaxel for standard of 6 cycles, and may be continued at the discretion of investigators. If the subject experiences progression, an unacceptable toxicity related to paclitaxel, or termination of lapatinib therapy, paclitaxel therapy must be terminated any time of study period, even before 6 cycles of paclitaxel are given.

This study consists of the Phase I and Phase II parts:

Phase I part

Tolerability and pharmacokinetics in 6 subjects will be evaluated in Phase I part of study and the tolerability criteria are set as follow:

Tolerability criteria in first cycle; Concerning the safety tolerability of this trial, if 1 out of 6 first enrolled subjects meets the tolerability criteria, the study will proceed to phase II part and the regimen will judged as well tolerable. If 2 subjects meet the tolerability criteria, the sponsor will consult the safety review committee. GSK will finally judge based on the consultation regarding the tolerability and the medical significance.

Grade 4 hematologic toxicities. Thrombocytopenia less than or equal to 25,000/mm3 Grade 3 or 4 and clinically significant non-haematologic toxicities. Inability to start cycle 2 within 2 weeks of scheduled dosing due to unresolved toxicity.

For all 6 subjects enrolled, safety profiles occurred in cycle 1 are closely monitored individually. When considering the appropriateness of study continuation, not only the safety profiles noted in cycle 1 of this study, but also the safety profiles reported from pilot part of EGF104578 study and other relevant studies will be referred in order to make medical decisions.

Phase II part After tolerability in 6 subjects enrolled in Phase I part is confirmed, further 6 subjects to be enrolled for Phase II part (i.e. total of 12 subjects). Subjects will receive a daily dose of lapatinib until disease progression or withdrawal from study treatment due to unacceptable toxicity or withdrawal of consent. All 12 subjects will be followed for survival.

ELIGIBILITY:
Inclusion Criteria:

* Prior written consent in participating in the study by the subject or his/her private attorney.
* Japanese female >=18 years of age.
* Invasive breast cancer with stage IV disease.
* Documentation by local laboratory of ErbB2 status by immunohistochemistry (IHC) or amplification by fluorescence in situ hybridization (FISH).
* If a taxane had been administered in the neoadjuvant or adjuvant setting, progression must have occurred >12 months after completion of this treatment and the patients recovered from all associated toxicities.
* Measurable lesion(s) according to RECIST criteria.
* Radiotherapy as palliative treatment for painful metastatic disease is permitted but must have been stopped within 2 weeks prior to initiation of any investigational treatment.
* For those patients whose disease is ER+ and/or PR+ one of the following criteria should be met:

  * Patient with visceral disease that requires chemotherapy (e.g., patients with liver or lung metastases).
  * Rapidly progressing or life threatening disease that are considered to be inapplicable to hormonal therapy, as determined by the investigator.
  * Patients who received hormonal therapy and are no longer benefiting from this therapy and the hormonal treatment must have been stopped before the first dose of investigational treatment.
  * Subjects recovered from all the associated toxicities by prior endocrine therapy.
* Eastern cooperative oncology group (ECOG) Performance status (PS) of 0 or 1.
* Able to swallow and retain oral medication.
* Cardiac ejection fraction within institutional range of normal as measured by echocardiogram. MUGA scan is accepted in cases where an echocardiogram cannot be performed or is inconclusive.
* Adequate organ function.

Exclusion Criteria:

* Pregnant or lactating females at anytime during the study.
* Received prior chemotherapy, immunotherapy, biologic therapy or anti-ErbB1/ErbB2 therapy for metastatic disease.
* History of other malignancy.
* Prior therapy with an ErbB1 and/or ErbB2 inhibitor, other than trastuzumab, in the adjuvant setting.
* Planned concurrent anti-cancer therapy (chemotherapy, radiation therapy, immunotherapy, biologic therapy, hormonal therapy) while taking investigational treatment.
* Used an investigational drug within 30 days or five half-lives, whichever is longer, preceding the first dose of investigational treatment.
* Unresolved or unstable, serious toxicity from prior administration of another investigational drug and/or of prior anti-cancer treatment.
* Uncontrolled infection.
* Patients having at least positive antibody either to HBs or HBc.
* Patients who have had a positive HCV antibody.
* Peripheral neuropathy grade 2 or greater.
* Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel. Subjects with ulcerative colitis are also excluded.
* Dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent.
* Known history or clinical evidence of central nervous system (CNS) metastases or leptomeningeal carcinomatosis.
* Concurrent disease or condition that would make the subject inappropriate for study participation or any serious medical disorder that would interfere with the subject's safety.
* Known history or concurrent condition of uncontrolled or symptomatic angina, arrhythmias, or congestive heart failure.
* Concurrent treatment with prohibited medications.
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to paclitaxel or lapatinib or their excipients.
* Have current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-04; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (8):
- Japan (8):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Ehime
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Kagoshima
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Saitama
  - GSK Investigational Site, Tokyo

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Six participants who met the eligibility criteria were enrolled into Phase I of the study. These 6 participants continued treatment into Phase II of the study, into which an additional 6 participants were enrolled. A total of 12 participants were followed until death or withdrawal from the study.
Groups:
- Lapatinib 1500 mg + Paclitaxel 80 mg/m^2: Participants received lapatinib 1500 milligrams (mg) once daily (QD) in combination with intravenous (IV) paclitaxel (80 milligrams per meters squared [mg/m^2]) weekly on Day 1, Day 8, and Day 15 of a 4-week cycle until disease progression or withdrawal from study treatment due to unacceptable toxicity or withdrawal of consent.
Period: Overall Study
Arm/Group | Lapatinib 1500 mg + Paclitaxel 80 mg/m^2
Started | 12
Completed | 6
Not Completed | 6
Not completed — Withdrawal due to death | 6

BASELINE CHARACTERISTICS:
Groups:
- Lapatinib 1500mg + Paclitaxel 80mg/m^2: Participants received lapatinib 1500 mg QD in combination with IV paclitaxel 80 mg/m^2 weekly on Day 1, Day 8, and Day 15 of a 4-week cycle until disease progression or withdrawal from study treatment due to unacceptable toxicity or withdrawal of consent.
Arm/Group | Lapatinib 1500mg + Paclitaxel 80mg/m^2
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.1 (7.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian - Japanese Heritage | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Intolerable Toxicities in Phase I of the Study
Description: Investigational treatment was considered tolerable if one or more of the tolerability criteria were met by none or one of the 6 participants in the first cycle of Phase I. If one or more tolerability criteria were met by two or more participants, the issue was referred to the safety committee. Tolerability criteria for toxicities related to investigational treatment included grade 4 neutropenia persisting for 7 or more days, thrombocytopenia with a platelet count of less than or equal to 25,000/millimeter (mm)^3 , clinically significant Grade 3 or 4 non-haematologic toxicities (excluding nausea) and inability to start cycle 2 within 2 weeks of scheduled dosing due to unresolved toxicity.
Time Frame: 28 days
Population: All Subjects Population: all participants who received at least one dose of study medication and participated in Phase I of the study.
Measure: Number; unit: Participants
Groups:
- Lapatinib 1500 mg + Paclitaxel 80 mg/m^2: Participants received lapatinib 1500 mg QD in combination with IV paclitaxel 80 mg/m^2 weekly on Day 1, Day 8, and Day 15 of a 4-week cycle until disease progression or withdrawal from study treatment due to unacceptable toxicity or withdrawal of consent.
Arm/Group | Lapatinib 1500 mg + Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 6
Participants | 1

2. Primary Outcome: Overall Survival
Description: Overall survival is defined as the time from the start of treatment until death due to any cause. For participants who survived, time to death was censored at the time of the last confirmation of survival.
Time Frame: From the start of treatment until death due to any cause or study close, whichever occurred first (assessed up to a maximum of 1290 Days)
Population: All Subjects Population: all participants who received at least one dose of study medication
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lapatinib 1500 mg + Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 12
Months | 35.6 [23.9 to NA] — Due to an insufficient number of events the upper limit of the 95% confidence Interval could not be calculated.

3. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the interval between the start of treatment and the earliest date of radiological disease progression or death due to any cause, whichever occurred first. PFS was based on the investigator's assessment. For participants who survived, time to death was censored at the time of the last confirmation of survival.
Time Frame: From the start of treatment until the earliest date of radiological disease progression or death due to any cause, whichever occured first (up to 1009 Days).
Population: All Subjects Population. Participants who met the following criteria were censored: no Baseline assessment, no progression, treatment discontinuation for undocumented progression, treatment discontinuation for toxicity or other reason, new anti-cancer treatment started, and death or progression after more than one missed visit.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lapatinib 1500 mg + Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 12
Months | 13.9 [7.6 to 27.9]

4. Secondary Outcome: Time to Response
Description: Time to response is defined as the time from the start of treatment until first documented evidence of partial response (PR) or a complete response (CR) (whichever status is recorded first). Analysis was based on responses confirmed at a repeat assessment made at least 4 weeks after the initial response, with the time to response taken as the first time the response was observed. CR is defined as the disappearance of all target lesions (TLs) and non-TLs. PR is defined as at least a 30% decrease in the sum of the longest diameter (LD) of the target lesions, taking as a reference, the Baseline sum LD. Baseline measurements were obtained at the Screening Visit.
Time Frame: From the start of treatment until the first documented evidence of a PR or CR, whichever status is recorded first (up to 66 Days).
Population: All Subjects Population. Only those participants with a CR or a PR were assessed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lapatinib 1500 mg + Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 10
Months | 1.9 [1.8 to 1.9]

5. Secondary Outcome: Duration of Response
Description: Duration of response is defined as the time from the first documented evidence of a CR or a PR until the first documented sign of disease progression or death due to any cause (whichever occured earlier). The analysis was based on responses as evaluated by the investigator and was confirmed at a repeat assessment, with the duration of response taken from the first time the response was observed. CR is defined as the disappearance of all TLs and non-TLs. PR is defined as at least a 30% decrease in the sum of the LD of the target lesions, taking as a reference, the Baseline sum LD. Baseline measurements were obtained at the Screening Visit.
Time Frame: From the first documented evidence of a CR or a PR until the first documented sign of disease progression or death, whichever occurred earlier (up to 953 Days).
Population: All Subjects Population. Only those participants with a CR or a PR were assessed. For participants who did not progress or die, duration of response was censored on the date of the last assessment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lapatinib 1500 mg + Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 10
Months | 14.5 [9.1 to 26.3]

6. Secondary Outcome: Number of Partcipants With a Best Overall Response (OR) as Determined by the Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Best OR was defined as the best response recorded from the start of treatment until progressive disease (PD)/death as assessed by the investigator. CR is defined as the disappearance of all TLs and non-TLs. PR is defined as at least a 30% decrease in the sum of the LD of the target lesions, taking as a reference, the Baseline sum LD. Baseline measurements were obtained at the Screening Visit. PD is defined as at least a 20% increase in the sum of the LD of target lesions or the appearance of 1 or more new lesions compared to the smallest sum LD recorded since the treatment started. Stable disease (SD) is defined as neither sufficient shrinkage to qualify for a PR nor sufficient increase to qualify for PD compared to the smallest sum LD since the treatment started. Any participant who could not be classified by the four preceding definitions was considered Not evaluable.
Time Frame: From the start of treatment until progressive disease/death (up to 1009 Days).
Population: All Subjects Population. All participants who received at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Lapatinib 1500 mg + Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 12
Participants
  CR | 0
  PR | 10
  SD | 1
  PD | 1
  Not evaluable | 0
  Unkown | 0

7. Secondary Outcome: Number of Participants With Clinical Benefit Response (CBR)
Description: CBR is defined using RECIST as the number of participants who received at least one dose of study medication and achieved a best OR classified as CR, PR or SD for at least 6 months (24 weeks), i.e., CR + PR + SD for >=24 weeks. CBR was based on confirmed responses by the investigator. CR is defined as the disappearance of all TLs and non-TLs. PR is defined as at least a 30% decrease in the sum of the LD of the target lesions, taking as a reference, the Baseline sum LD. Baseline measurements were obtained at the Screening Visit. PD is defined as at least a 20% increase in the sum of the LD of TLs or the appearance of 1 or more new lesions compared to the smallest sum LD recorded since the treatment started. SD is defined as neither sufficient shrinkage to qualify for a PR nor sufficient increase to qualify for PD compared to the smallest sum LD since the treatment started. Any participant who could not be classified by the the four preceding definitions was considered Not evaluable
Time Frame: From the start of treatment until progressive disease/death (up to 1009 Days).
Population: All Subjects Population. All participants who received at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Lapatinib 1500 mg + Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 12
Participants
  Complete response | 0
  Partial response | 10
  Stable disease >=24 weeks | 0
  Stable disease <=24 weeks | 1
  Progressive disease | 1
  Not evaluable | 0
  Unknown | 0

8. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Lapatinib and Paclitaxel
Description: Cmax is defined as the maximum concentration of lapatinib and paclitaxel. Cmax was calculated from lapatinib plasma concentration-time data on Day 8 and Day 14 and paclitaxel plasma concentration-time data on Day 1 and Day 8 with model-independent analyses
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post-dose on Day 8 and Day 14 for lapatininb; Day 1 and Day 8 for paclitaxel
Population: Pharmacokinetic (PK) Population: all participants who provided blood samples for PK evaluation
Measure: Geometric Mean (95% Confidence Interval); unit: Nanogram per milliliter ng/mL
Arm/Group | Lapatinib 1500 mg + Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 6
Nanogram per milliliter ng/mL
  Lapatinib 1500 mg, Day 14 | 5945.022 [3077.881 to 11482.989]
  Lapatinib 1500 mg +Paclitaxel 80 mg/m^2, Day 8 | 9470.401 [7157.899 to 12530.003]
  Paclitaxel 80 mg/m^2, Day 1 | 3485.229 [2693.037 to 4510.455]
  Paclitaxel 80 mg/m2+ Lapatinib 1500 mg, Day 8 | 3412.332 [2753.083 to 4229.443]

9. Secondary Outcome: Area Under the Concentration-time Curve (AUC) (0-24) of Lapatinib and Paclitaxel
Description: AUC is defined as the area under the lapatinib or paclitaxel concentration-time curve from time 0 to 24 hours (hrs). AUC (0-24) was calculated from lapatinib plasma concentration-time data on Day 8 and Day 14 and paclitaxel plasma concentration-time data on Day 1 and Day 8 with model-independent analyses
Time Frame: as for outcome 8
Population: PK Population: all participants who provided blood samples for PK evaluation
Measure: Geometric Mean (95% Confidence Interval); unit: hours * nanograms/milliliter (hr*ng/mL)
Arm/Group | Lapatinib 1500 mg + Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 6
hours * nanograms/milliliter (hr*ng/mL)
  Lapatinib 1500 mg, Day 14 | 79518.047 [34664.607 to 182408.525]
  Lapatinib 1500 mg + Paclitaxel 80 mg/m^2, Day 8 | 113078.292 [74630.131 to 171334.285]
  Paclitaxel 80 mg/m^2, Day 1 | 4657.218 [3942.630 to 5501.322]
  Paclitaxel 80mg/m^2 + Lapatinib 1500 mg, Day 8 | 5786.123 [4667.500 to 7172.837]

10. Secondary Outcome: AUC From Time Zero to Infinity (0-INF) of Paclitaxel
Description: AUC(0-INF) is area under the plasma concentration-time curve from time 0 extrapolated to infinity. AUC (0-INF) was calculated from paclitaxel plasma concentration-time data on Day 1 and Day 8 with model-independent analyses
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post-dose on Day 1 and Day 8 for paclitaxel
Population: PK Population: all participants who provided blood samples for PK evaluation
Measure: Geometric Mean (95% Confidence Interval); unit: hr*ng/mL
Arm/Group | Lapatinib 1500 mg + Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 6
hr*ng/mL
  Paclitaxel 80 mg/m^2, Day 1 | 5125.908 [4371.289 to 6010.798]
  Paclitaxel 80mg/m^2 + Lapatinib 1500 mg, Day 8 | 6279.964 [5005.596 to 7878.773]

11. Secondary Outcome: Time to the Maximum Drug Concentration (Tmax) of Lapatinib and Paclitaxel
Description: Tmax is defined as the time to peak concentration from initiation of lapatinib and paclitaxel dosing. Tmax was calculated from lapatinib plasma concentration-time data on Day 8 and Day 14 and paclitaxel plasma concentration-time data on Day 1 and Day 8 with model-independent analyses
Time Frame: as for outcome 8
Population: PK Population: all participants who provided blood samples for PK evaluation
Measure: Median (Full Range); unit: Hr
Arm/Group | Lapatinib 1500 mg + Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 6
Hr
  Lapatinib 1500 mg, Day 14 | 4.992 [1.50 to 6.08]
  Lapatinib 1500 mg + Paclitaxel 80 mg/m^2, Day 8 | 4.975 [1.95 to 6.00]
  Paclitaxel 80 mg/m^2, Day 1 | 0.992 [0.95 to 1.08]
  Paclitaxel 80mg/m^2 + Lapatinib 1500 mg, Day 8 | 0.975 [0.50 to 1.02]

12. Secondary Outcome: Distribution Volume at Steady State (Vss) of Paclitaxel
Description: Vss is the volume of distribution at steady state of paclitaxel. Vss was calculated from paclitaxel plasma concentration-time data on Day 1 and Day 8 with model-independent analyses
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post-dose on Day 1 and Day 8 for paclitaxel
Population: PK Population: all participants who provided blood samples for PK evaluation
Measure: Geometric Mean (95% Confidence Interval); unit: milliliter per meters squared (mL/m^2)
Arm/Group | Lapatinib 1500 mg + Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 6
milliliter per meters squared (mL/m^2)
  Paclitaxel 80 mg/m^2, Day 1 | 98909.326 [73404.017 to 133276.831]
  Paclitaxel 80mg/m^2 + Lapatinib 1500 mg, Day 8 | 77460.104 [63942.340 to 93835.598]

13. Secondary Outcome: Half-life (t1/2) of Paclitaxel
Description: Half-life is defined as the time required for the amount of the drug in the plasma to decrease by half. T1/2 was calculated from paclitaxel plasma concentration-time data on Day 1 and Day 8 with model-independent analyses
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post-dose on Day 1 and Day 8 for paclitaxel
Population: PK Population: all participants who provided blood samples for PK evaluation
Measure: Geometric Mean (95% Confidence Interval); unit: Hr
Arm/Group | Lapatinib 1500 mg + Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 6
Hr
  Paclitaxel 80 mg/m^2, Day 1 | 12.186 [10.055 to 14.768]
  Paclitaxel 80mg/m^2 + Lapatinib 1500 mg, Day 8 | 9.855 [8.477 to 11.457]

14. Secondary Outcome: Drug Clearance (CL) of Paclitaxel
Description: CL is defined as the volume of plasma in the vascular compartment cleared of drug per unit time by the processes of metabolism and excretion. CL was calculated from paclitaxel plasma concentration-time data on Day 1 and Day 8 with model-independent analyses
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post-dose on Day 1 and Day 8 for paclitaxel
Population: PK Population: all participants who provided blood samples for PK evaluation.
Measure: Geometric Mean (95% Confidence Interval); unit: mL/hour/m^2
Arm/Group | Lapatinib 1500 mg + Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 6
mL/hour/m^2
  Paclitaxel 80 mg/m^2, Day 1 | 15606.990 [13309.380 to 18301.238]
  Paclitaxel 80mg/m^2 + Lapatinib 1500 mg, Day 8 | 12738.926 [10153.865 to 15982.114]

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the start of study medication until 30 days after the last dose (up to 1045 Days).
Description: SAEs and non-serious AEs are reported for members of the All Subjects Population, comprised of all participants who had received at least one dose of the study medication.
Arm/Group | Lapatinib 1500 mg + Paclitaxel 80 mg/m^2
Serious Adverse Events (participants affected / at risk) | 3/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lapatinib 1500 mg + Paclitaxel 80 mg/m^2 (N=12)
Neutrophil count decreased (Investigations) | 2
Left ventricular dysfunction (Cardiac disorders) | 1
Pneumonia (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lapatinib 1500 mg + Paclitaxel 80 mg/m^2 (N=12)
Diarrhoea (Gastrointestinal disorders) | 11
Stomatitis (Gastrointestinal disorders) | 8
Vomiting (Gastrointestinal disorders) | 6
Nausea (Gastrointestinal disorders) | 5
Abdominal pain upper (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 3
Cheilitis (Gastrointestinal disorders) | 2
Dental caries (Gastrointestinal disorders) | 2
Haemorrhoids (Gastrointestinal disorders) | 2
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Glossitis (Gastrointestinal disorders) | 1
Periproctitis (Gastrointestinal disorders) | 1
Proctalgia (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Haemoglobin decreased (Investigations) | 10
Alanine aminotransferase increased (Investigations) | 7
Aspartate aminotransferase increased (Investigations) | 6
Haematocrit decreased (Investigations) | 6
Blood alkaline phosphatase increased (Investigations) | 5
Weight decreased (Investigations) | 4
Blood albumin decreased (Investigations) | 3
Neutrophil count decreased (Investigations) | 3
White blood cell count decreased (Investigations) | 3
Basophil count decreased (Investigations) | 2
Blood bilirubin increased (Investigations) | 2
Monocyte count decreased (Investigations) | 2
Platelet count increased (Investigations) | 2
Red blood cell count decreased (Investigations) | 2
Blood glucose increased (Investigations) | 1
Blood potassium decreased (Investigations) | 1
Blood potassium increased (Investigations) | 1
Blood urea increased (Investigations) | 1
Electrocardiogram QT prolonged (Investigations) | 1
Eosinophil count decreased (Investigations) | 1
Neutrophil count increased (Investigations) | 1
White blood cell count increased (Investigations) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 12
Rash (Skin and subcutaneous tissue disorders) | 8
Nail disorder (Skin and subcutaneous tissue disorders) | 6
Dry skin (Skin and subcutaneous tissue disorders) | 2
Erythema (Skin and subcutaneous tissue disorders) | 2
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2
Acne (Skin and subcutaneous tissue disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1
Keratolysis exfoliativa acquired (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 8
Dysgeusia (Nervous system disorders) | 5
Headache (Nervous system disorders) | 2
Hypoaesthesia (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 8
Neutropenia (Blood and lymphatic system disorders) | 8
Lymphopenia (Blood and lymphatic system disorders) | 6
Erythropenia (Blood and lymphatic system disorders) | 3
Fatigue (General disorders) | 8
Oedema (General disorders) | 3
Oedema peripheral (General disorders) | 3
Pyrexia (General disorders) | 3
Mucosal inflammation (General disorders) | 2
Discomfort (General disorders) | 1
Feeling drunk (General disorders) | 1
Feeling hot (General disorders) | 1
Injection site reaction (General disorders) | 1
Malaise (General disorders) | 1
Paronychia (Infections and infestations) | 7
Nasopharyngitis (Infections and infestations) | 6
Gingivitis (Infections and infestations) | 2
Bronchitis (Infections and infestations) | 1
Cystitis (Infections and infestations) | 1
Erysipelas (Infections and infestations) | 1
Folliculitis (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Nail infection (Infections and infestations) | 1
Subcutaneous abscess (Infections and infestations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 7
Dehydration (Metabolism and nutrition disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 1
Blepharitis (Eye disorders) | 1
Cataract (Eye disorders) | 1
Erythema of eyelid (Eye disorders) | 1
Eyelid oedema (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Fractured coccyx (Injury, poisoning and procedural complications) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1
Vaginal discharge (Reproductive system and breast disorders) | 1
Vaginal inflammation (Reproductive system and breast disorders) | 1
Cardiomegaly (Cardiac disorders) | 1
Left ventricular dysfunction (Cardiac disorders) | 1
Meniere's disease (Ear and labyrinth disorders) | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Insomnia (Psychiatric disorders) | 1
Neurogenic bladder (Renal and urinary disorders) | 1
Hot flush (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.